CLINICAL TRIAL: NCT06541314
Title: A Multicenter, Single-Arm Clinical Study of Fluzoparib Monotherapy As Neoadjuvant Treatment for Advanced Epithelial Ovarian Cancer
Brief Title: Fluzoparib Neoadjuvant Therapy for Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202404-015-1
Record Dates: First submitted 2024-06-13; First posted 2024-08-07 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fluzoparib neoadjuvant therapy (Experimental)
  Interventions: Drug: Fluzoparib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib (50mg per capsule) 150mg po bid, with a treatment cycle of 28 days. Administer 2 cycles in total.

SUMMARY:
This study is an interventional, single-arm, open-label clinical trial. To evaluate the safety and efficacy of Fluzoparib as neoadjuvant therapy in patients with FIGO stage III and IV , BRCA mutations or HRD positive epithelial ovarian cancer who cannot achieve R0 surgery as assessed by imaging (Suidan's CT score) or laparoscopy (Fagotti score), or cannot tolerate surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years.
2. Biopsies obtained via open surgery, laparoscopic surgery, or needle biopsy, confirmed by professional pathologists as high-grade serous or endometrioid ovarian cancer, peritoneal cancer, or fallopian tube cancer (hereinafter referred to as ovarian cancer); FIGO stage III-IV.
3. Presence of BRCA1/2 mutation or HRD positivity confirmed in tissue or blood samples by the designated testing institution of the study center.
4. Before any trial procedures begin, an informed consent form must be signed according to the principle of informed consent and filed at the study center.
5. The patient must have at least one measurable lesion that can be assessed by CT or MRI (RECIST 1.1).
6. Blood and tissue samples from patients can be obtained before, during, and after treatment, and subjects agree to submit blood and tissue samples to the central laboratory for the purpose of expansion research for this trial, including but not limited to: (1) possible gene-related research; (2) Possible tumor marker-related research.
7. Patients deemed unable to achieve R0 cytoreduction or unable to tolerate surgery by gynecologic oncologists at the study center: (1) Fagotti laparoscopic score ≥ 8 points; (2) When laparoscopic assessment is difficult to perform, an upper abdominal CT score ≥ 3 points may be used. Criteria for determining inability to tolerate surgery may include: (1) BMI ≥ 40.0; (2) Multiple chronic diseases; (3) Malnutrition or hypoproteinemia; (4) Moderate to large amounts of ascites; (5) Newly diagnosed venous thromboembolism; (6) ECOG > 2.
8. Expected survival time > 12 weeks.
9. Patients with an ECOG score of 0-2.
10. Good organ function. (1) Bone marrow function: NEUT ≥ 1.5*10^9/L; PLT ≥ 100*10^9/L; HGB ≥ 100g/L. (2) Liver function: TBIL ≤ 1.5 times the upper limit of normal or DBIL ≤ 1.0 times the upper limit of normal; AST and ALT ≤ 2.5 times the upper limit of normal, and in the presence of liver metastasis, must be ≤ 5 times the upper limit of normal. (3) Renal function: serum creatinine ≤ 1.5 times the upper limit of normal, or creatinine clearance rate ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).
11. For women of reproductive age, a negative blood or urine pregnancy test within one week prior to enrollment is required, and effective contraceptive measures must be taken after enrollment, such as using physical barrier methods (condoms) or complete abstinence. The use of oral, injectable, or implantable hormonal contraceptives is not permitted. Or women who are not of reproductive age, defined as those who have naturally entered menopause and have been amenorrheic for over a year, have undergone surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy), or have serum follicle-stimulating hormone, luteinizing hormone, and plasma estradiol levels within the menopausal range as specified by the study center laboratory.
12. Understand the trial process and voluntarily sign the informed consent form, with the ability to comply with the trial protocol for the duration of the study, including cooperating with any required treatments, examinations, tests, follow-ups, and questionnaires.
13. Patients are willing to complete quality of life questionnaires during the trial treatment and follow-up process, and agree that the results of these questionnaires may be used for clinical research.
14. Any prior chemotherapy-related toxicities must have resolved to ≤ CTCAE grade 1 or baseline levels, except for stable grade 2 or lower sensory neuropathy or alopecia.

Exclusion Criteria:

1. Concurrent use of other investigational drugs or participation in other clinical drug trials during this study.
2. Concurrent use of other neoadjuvant treatments for cancer during this study, including but not limited to chemotherapy, radiotherapy, immunotherapy, microbial therapy, traditional Chinese medicine, and other experimental therapies.
3. Known allergy to Fluzoparib or any active or inactive components with a similar chemical structure to Fluzoparib.
4. Unable to swallow oral medications, and having any gastrointestinal disorders that may interfere with the absorption or metabolism of the study drug, such as uncontrolled nausea and vomiting, gastrointestinal obstruction, or malabsorption.
5. Received any cancer-related treatment for ovarian cancer.
6. Previously received known or potential PARP inhibitor therapy.
7. Symptomatic or uncontrollable brain metastases requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids, or clinical manifestations of spinal cord compression.
8. History of severe venous thrombosis or pulmonary embolism.
9. Received other molecular targeted therapy within 4 weeks before enrollment.
10. Symptomatic or uncontrollable brain metastases requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids, or clinical manifestations of spinal cord compression.
11. Undergone major surgery within 3 weeks before the start of the study, or not yet recovered from surgery.
12. Presence of uncorrected electrolyte disturbances at the time of dosing.
13. Subjects have had other malignant diseases in the past 3 years, except for effectively treated skin squamous cell carcinoma, basal cell carcinoma, ductal carcinoma in situ of the breast, or cervical carcinoma in situ.
14. Patients have a history of or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
15. Patients with severe, uncontrolled diseases or whom the investigator judges to be generally unsuitable for inclusion in the study, including but not limited to: active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.; severe cardiovascular diseases, uncontrolled ventricular arrhythmias, myocardial infarction within the last 3 months; uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental disorders that may affect the patient's ability to sign the informed consent; uncontrolled hypertension; immunodeficiency (excluding splenectomy) or other conditions that the investigator considers may expose the patient to high-risk toxicity.
16. Any medical history or existing clinical evidence suggesting potential confounding of study results, interference with patient compliance with the study protocol throughout the study treatment period, or not in the best interest of the patient.
17. The patient received a platelet or red blood cell transfusion within 3 days before the start of treatment with the study drug.
18. Pregnant or lactating patients, or those planning to become pregnant during the study treatment period.
19. Clinically unresolved prior treatment toxicity (≥ grade 2), excluding alopecia, neuropathy, lymphocytopenia, and skin hypopigmentation.
20. Persons involved in the planning or implementation of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
ORR | From the diagnosis of epithelial ovarian cancer until the completion of neoadjuvant monotherapy with Fluzoparib, assessed up to 10 weeks.
  Objective response rate. After completing neoadjuvant monotherapy with Fluzoparib, the proportion of patients who achieve complete response and partial response according to the RECIST 1.1 criteria.
R0 Resection Rate | From the completion neoadjuvant monotherapy with Fluzoparib until the date of surgery, with the assessment of R0 resection rate occurring within 1 to 2 weeks after treatment completion.
  To evaluate the proportion of patients with advanced epithelial ovarian cancer, initially deemed non-R0 resectable or unable to tolerate surgery, who achieve R0 resection following neoadjuvant monotherapy with Fluzoparib.

SECONDARY OUTCOMES:
PFS | The time from patient enrollment until the date of first documented tumor progression or death from any cause, whichever occurs first, assessed up to 60 months.
  Progression-free survival. The time from patient enrollment to tumor progression or death.
OS | From the time from patient enrollment until the date of death from any cause, assessed up to 120 months.
  Overall survival. The time from patient enrollment to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China